CLINICAL TRIAL: NCT00685568
Title: Phase I Pilot Toxicity/Methods Validation Study of Celecoxib in Genotype-Positive Children With Familial Adenomatous Polyposis
Brief Title: Celecoxib in Preventing Colorectal Cancer in Young Patients With a Genetic Predisposition for Familial Adenomatous Polyposis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ID02-090; MDA-ID-02090; CDR0000596468 (Other: NCI Clinical Trials)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Cancer; Precancerous Condition
Keywords: colon cancer; rectal cancer; familial adenomatous polyposis
MeSH Terms: conditions — Colorectal Neoplasms; Precancerous Conditions; Colonic Neoplasms; Rectal Neoplasms; Adenomatous Polyposis Coli | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral celecoxib twice daily for 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: celecoxib
- Arm II (Placebo Comparator): Patients receive oral placebo twice daily for 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: celecoxib — Orally, twice daily for 3 months; 50 mg tablets. Celecoxib escalating doses starting at 4 mg/kg/day.
  Arms: Arm I
Other: placebo — Orally, twice daily for 3 months
  Arms: Arm II

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of celecoxib may keep polyps and colorectal cancer from forming in patients with familial adenomatous polyposis.

PURPOSE: This randomized phase I trial is studying the side effects and best dose of celecoxib in treating young patients with a genetic predisposition for familial adenomatous polyposis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and toxicity of celecoxib in pediatric patients with genotype-positive familial adenomatous polyposis.

Secondary

* Determine the aberrant crypt foci (ACF) and adenoma burden in the entire colorectum of these patients.
* Eliminate the learning curve in a phase II/III trial (reproducibility of endoscopic techniques, tolerability of procedure).
* Compare sedation strategies based on local standards (monitored anesthesia care vs conscious sedation).
* Validate the ACF scoring technique.
* Establish the short-term (3 month) impact of celecoxib on ACF count in order to determine appropriateness of ACF as a pathologic endpoint in a phase II/III trial.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral celecoxib twice daily for 3 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo twice daily for 3 months in the absence of disease progression or unacceptable toxicity.

Patients undergo colonoscopy at baseline and at 3 months. Patients also complete psychosocial questionnaires at baseline.

Blood samples are collected at baseline to assess the influence of polymorphisms (CYP2C9, uridine diphosphate (UDP)-glucuronosyl transferase, A6, glutathione S-transferase [GST] M1, and Glutathione S-transferase (GST) theta 1 (GSTT1)) on age of onset of phenotype or number of colorectal polyps. Plasma drug trough levels are assessed at baseline, 1 month, and 3 months.

After completion of study treatment, patients are followed periodically for up to 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of familial adenomatous polyposis (FAP) based on genetic predisposition testing
* Genotype-positive FAP (pathologic Adenomatous polyposis coli (APC) mutation)

  * No attenuated FAP genotype, defined by any of the following:

    * Mutation at the 5' end of APC and exon 4
    * Exon 9-associated phenotypes
    * 3' region mutations
* Has an intact colon

  * No requirement for colectomy
  * Parent(s) do not desire colectomy (regardless of adenoma burden)
* Colorectal adenoma burden as assessed by baseline colonoscopy

  * No diagnosis of severe dysplasia or greater
  * No more than 10 adenomas ≥ 1 cm
  * No more than 100 adenomas of any size
  * No evidence of anemia (hematocrit < 33%)
* No new diagnosis of carcinoma

PATIENT CHARACTERISTICS:

* White Blood Count (WBC) > 3,000/μL
* Platelet count > 100,000/μL
* Hemoglobin > 10.0 g/dL
* Aspartate aminotransferase/alanine aminotransferase (AST/ALT) < 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 1.5 times ULN
* Total bilirubin < 1.5 times ULN
* Creatinine < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of hypersensitivity to COX-2 inhibitors, sulfonamides, NSAIDs, or salicylates
* No history of peptic ulcer disease
* No significant medical or psychiatric problem that, in the opinion of the principal investigator, would make the patient a poor candidate for the study
* No other unacceptable clinical risk (e.g., previously unknown bleeding diatheses)
* No invasive carcinoma within the past 5 years

PRIOR CONCURRENT THERAPY:

* More than 3 months since prior investigational agent
* More than 6 months since prior chemotherapy
* No prior radiotherapy to the pelvis
* At least 3 months since prior NSAIDs (at any dose) at a frequency of ≥ 3 times/week
* At least 1 month since prior NSAIDs (at any dose) at a frequency of < 3 times/week
* At least 1 month since prior nasal steroids
* Concurrent Nonsteroidal Antiinflammatory Drugs (NSAIDs) allowed provided they are administered ≤ 5 times per month
* Concurrent orally inhaled steroids allowed provided they are administered for ≤ 4 weeks over a 6-month period
* Concurrent oral or intravenous (IV) corticosteroids allowed provided they are administered for ≤ 2 consecutive weeks over a 6-month period
* Concurrent proton pump inhibitors to treat gastric reflux allowed
* No concurrent nasal steroids except mometasone (Nasonex)
* No concurrent fluconazole, lithium, or adrenocorticosteroids

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2002-11-21 (Actual); Primary Completion 2006-04-21 (Actual); Study Completion 2006-04-21 (Actual)

PRIMARY OUTCOMES:
Toxicity | 3 months

SECONDARY OUTCOMES:
Aberrant crypt foci (ACF) and adenoma burden in the entire colorectum | 3 months
Elimination of the learning curve in a phase II/III trial | 3 months
Comparison of sedation strategies based on local standards | 3 months
Validation of technique for scoring ACFs | 3 months
Short-term (3 month) impact of celecoxib on ACF count | 3 months
Adherence | 3 months
Influence of polymorphisms on age of onset of phenotype or on the number of colorectal polyps | 3 months
Feasibility of psychosocial questionnaires | 3 months
Pharmacokinetics (plasma drug trough concentrations) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M. Lynch, MD, JD, Study Chair — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Medical School at Houston, Houston, Texas

REFERENCES:
- [Result] Lynch PM, Ayers GD, Hawk E, Richmond E, Eagle C, Woloj M, Church J, Hasson H, Patterson S, Half E, Burke CA. The safety and efficacy of celecoxib in children with familial adenomatous polyposis. Am J Gastroenterol. 2010 Jun;105(6):1437-43. doi: 10.1038/ajg.2009.758. Epub 2010 Mar 16. PMID 20234350